CLINICAL TRIAL: NCT06009822
Title: Investigation of Kinesiophobia and Functional Status of Patients After MPFL Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Research asistant (PT), Gazi University
Other Study IDs: Iayas4
Record Dates: First submitted 2023-08-08; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Medial Patellofemoral Dislocation; Kinesiophobia
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Medial Patellofemoral Ligament reconstruction: Must have undergone unilateral medial patellofemoral ligament (MPFL) reconstruction.
  At least 2 years post MPFL reconstruction surgery. Absence of patellar instability subsequent to the surgical procedure. Exclusion of patients with any orthopedic or neurological issues that might impact functionality, except for those who have undergone unilateral MPFL reconstruction.
  Interventions: Other: Postoperative outcome measurements

INTERVENTIONS:
Other: Postoperative outcome measurements — Kinesiophobia; It will be assessed on the Tampa Kinesiophobia Scale. Function; Lysholm knee score, kujala knee score, single-leg hop test, Y balance test and single leg sway index will be evaluated.
  Biodex Bio-balance system device will be used for single leg sway index.

SUMMARY:
Our aim in this study is to examine the functional and clinical results of patients who have undergone MPFL reconstruction at least 2 years after the operation. The presence of kinesiophobia of the patients will be evaluated and its relationship with functional outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Undergone unilateral medial patellofemoral ligament (MPFL) reconstruction
* At least 2 years after the operation

Exclusion Criteria:

* Patellar instability
* Knee ligament injury
* Meniscus injury
* Knee osteoarthritis
* Ankle ligament injury
* Ankle osteoarthritis
* Any neurological disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent unilateral MPFL reconstruction in the Department of Orthopedics and Traumatology, Gazi University Hospital between 2004 and 2019
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | up to 3 months
  Kinesiophobia refers to an excessive, irrational fear of movement or physical activity. The Tampa Scale for Kinesiophobia was used for assessment. The Tampa Scale for Kinesiophobia is scored between 17-68. A high score indicates high kinesiophobia.

SECONDARY OUTCOMES:
Knee Score | up to 3 months
  Function will be measured by the Lysholm knee score.The total score on the Lysholm Knee Score questionnaire can range from 0 to 100, with higher scores indicating better knee function and less impairment. General breakdown of the score interpretation:
  95-100: Excellent knee function 84-94: Good knee function 65-83: Fair knee function Below 65: Poor knee function
Patellofemoral Knee Score | up to 3 months
  Function will be measured by the Kujala Patellofemoral Knee Score. The total score on the Kujala Patellofemoral Knee Score questionnaire can range from 0 to 100, with higher scores indicating better knee function and less impairment. General breakdown of the score interpretation:
  100: No limitations or symptoms 85-99: Mild limitations or symptoms 70-84: Moderate limitations or symptoms Below 70: Severe limitations or symptoms
Single-leg hop test | up to 3 months
  The single-leg hop distance is an indicator of lower extremity function. The test evaluates an individual's lower limb strength, power, and overall functional performance. It specifically focuses on assessing an individual's ability to generate power and stability while performing a single-leg hop for maximal distance. When performing the test, the individual starts by standing on one leg at the starting point. The opposite leg is lifted slightly off the ground, and the hands can be placed on the hips or kept at the sides for balance. On the command to start, the individual hops forward on the single leg, aiming to jump as far as possible while maintaining control and balance. Perform 3 repetitions and record the longest distance jumped.
Dynamic balance | up to 3 months
  Dynamic balance will be measured by Y Balance Test. The Y Balance Test involves a person standing on one leg while reaching in anterior (forward), posteromedial (backward and to the side), and posterolateral (backward and to the other side) directions with the other leg. The person places their stance foot at the starting point on the central part of the Y-shaped device.While maintaining balance on the stance leg, the person reaches the free leg as far as possible along each of the three arms of the Y.The distance reached in each direction is measured and recorded.
Static balance | up to 3 months
  Static balance will be measured using a Biodex Balance System, single leg sway index test procedure. The device reports the person's body oscillations as sway index. A high stability index indicates poor postural control.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Hazar, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.